CLINICAL TRIAL: NCT03368976
Title: Prospective, Multicenter, Single Arm Feasibility Study to Collect Patient and Imaging Data for Avanos Medical Ultrasound Guided Regional Anesthesia System Development
Brief Title: PACMAN Ultrasound Recording Data Collection
Status: Terminated | Type: Observational
Why Stopped: Interim Goals met. Decision made to terminate in favor of completing the study as a second protocol in the future.
Sponsor: Avanos Medical (Other)
Responsible Party: Sponsor
Other Study IDs: 101-17-0001
Record Dates: First submitted 2017-12-06; First posted 2017-12-11 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Anesthesia, Local

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Interscalene
- Supraclavicular
- Infraclavicular
- Transversus Abdominus Plane
- Paravertebral Space
- Fascia Iliaca
- Femoral Nerve
- Saphenous Nerve via Adductor Canal
- Popliteal Sciatic Nerve

SUMMARY:
Study to collect videos of ultrasound recordings during peripheral nerve block procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older with underlying pathologies requiring surgical intervention facilitated by a specific regional nerve block
* Informed consent executed

Exclusion Criteria:

* Patients unable to understand and provide written consent
* Infection at the injection site
* Allergy to local anesthetic agents
* Medical condition obscuring visualization
* Known neuropathy at or around target nerve for the PNB
* Inability to communicate with the investigator or hospital staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with planned peripheral nerve block procedures.
Sampling Method: Non-Probability Sample
Enrollment: 767 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Collection of ultrasound recordings | 6 months
  Collection of 100 ultrasound recordings for each group

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - George Washington University, Washington D.C., District of Columbia
  - Andrews Institute, Gulf Breeze, Florida
  - University of Miami, Miami, Florida
  - Indiana University, Indianapolis, Indiana
  - Universal Medical Resources, Troy, Michigan
  - University of Minnesota - Twin Cities, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - Christ Hospital, Cincinnati, Ohio